CLINICAL TRIAL: NCT00273494
Title: Scandinavian Neoadjuvant Phase III Study of Induction Chemotherapy Followed by Irradiation Alone or Surgery Plus Irradiation in NSCLC Stage IIIA/N2 (T1N2, T2N2, T3/N2).
Brief Title: Neoadjuvant Chemotherapy Plus/Minus Surgery in Non-Small-Cell Lung Cancer (NSCLC) Stage IIIA/N2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Surgery in NSCLC stage IIIA/N2
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: N2 disease; Non-small cell lung cancer; Surgery; Neoadjuvant chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Procedure: Surgery

SUMMARY:
Hypothesis is that surgery is of benefit in locally advanced NSCLC with N2 disease.

Patients are randomised to surgery or not.

DETAILED DESCRIPTION:
Patients are after staging randomised to neoadj. chemotherapy followed by surgery followed by irradiation or to chemotherapy followed by irradiation.

Endpoint is survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified NSCLC
* Stage IIIA/N2
* age 18-75
* Lung function test allowing surgery
* Mediastinoscopy performed

Exclusion Criteria:

* Prior chemotherapy
* Prior irradiation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 1998-01; Study Completion 2008-01

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Jens B. Sorensen, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Dept. Oncology, Rigshospitalet, Copenhagen, Copenhagen, Denmark